CLINICAL TRIAL: NCT06580782
Title: Calcium Carbonate to Augment Labor Contractions
Acronym: CALC
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 24-07027775
Record Dates: First submitted 2024-08-28; First posted 2024-08-30 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Labor Dystocia; Labor Induction; Labor Augmentation
Keywords: Labor; Pregnancy; Labor Augmentation; Calcium Carbonate; labor induction
MeSH Terms: conditions — Dystocia | interventions — Calcium Carbonate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Data Analyst will be masked to the interventions assigned to participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Pitocin (Active Comparator): Control group will receive only the standard-dose synthetic oxytocin (Pitocin) alone for labor induction or augmentation.
  Interventions: Drug: Standard Dose Synthetic Pitocin
- Calcium Carbonate with Pitocin (Experimental): Participants will start an oral calcium carbonate regimen at the same time as initiating synthetic oxytocin (Pitocin) infusion.
  Interventions: Drug: Calcium Carbonate 500 MG; Drug: Standard Dose Synthetic Pitocin

INTERVENTIONS:
Drug: Calcium Carbonate 500 MG — Calcium Carbonate 500mg, orally, every 4 hours.
  Arms: Calcium Carbonate with Pitocin
Drug: Standard Dose Synthetic Pitocin — The participant will receive thestandard-dose synthetic oxytocin for labor induction or augmentation.

SUMMARY:
The investigators think that calcium carbonate can act as an assistive medication to improve contractions during labor.

DETAILED DESCRIPTION:
This study plans to study the acceptance and safety of using calcium carbonate as an medicine to help the labor induction process. The study aims to find if the use of calcium carbonate will lead to better labor contractions and increase the percentage of vaginal deliveries and improve delivery outcomes.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Nulliparas (no prior pregnancy lasting 20 weeks or greater of gestation)
* Gestational age above 36 weeks, at enrollment
* Present for induction or augmentation of labor inclusive of medical indication, elective induction at greater than 39 weeks' gestation, trial of labor after cesarean
* Singleton gestation (a multiple gestation reduced to a singleton, either spontaneously or therapeutically, before 14 0/7 weeks of gestation is acceptable)
* Ability to give informed consent
* Planned to undergo initiation of oxytocin infusion by their maternity care provider

Exclusion Criteria:

* Unable to understand or read English
* Presence of tachysystole (defined as more than 5 contractions in 10 minutes averaged over 30 minutes), recurrent variable or late fetal decelerations, and bradycardia in the prior 30 minutes before enrollment
* Non-vertex presenting fetus at enrollment
* Planned for cesarean delivery or contraindication to labor by institutional policy (e.g., placenta previa, vasa previa, active genital herpes infection, previous transmural myomectomy)
* Multi-fetal gestation (twins, triplets, and higher order multiples)
* Known contraindication to taking calcium carbonate including renal calculus, high urine calcium levels, elevated serum calcium, low serum phosphate, achlorhydria, or suspected digoxin toxicity.
* Deliveries with fetal chronic and/or pregnancy-related conditions, IUFD (Intra Uterine Fetal Death) or premature < 36 weeks of gestation.
* Major fetal anomaly suspected prenatally (defined as a fetal anomaly with anticipated neonatal intensive care unit admission)
* Suspected alloimmunization (given the increased likelihood for anticipated neonatal intensive care unit admission)
* Known severe fetal growth restriction (estimated fetal weight <3rd percentile) or abnormal umbilical artery Doppler studies (given the increased likelihood for anticipated neonatal intensive care unit admission)
* Participation in another interventional study that influences management of labor and delivery or perinatal morbidity or mortality
* Known allergic reactions to synthetic oxytocin intravenous solution or to Calcium Carbonate
* Significantly impaired consciousness or executive function (e.g., intubated or sedated)
* Patients treated with calcium channel blockers such as nifedipine or magnesium.
* Chronic renal failure and hyperphosphatemia.
* Inability to tolerate oral intake (i.e., nausea/vomiting)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-11-18 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Consented | Day 0
  RedCAP is used to track the consent rates to determine the feasibility of a larger randomized controlled trial.
Number of Participants Enrolled | Day 0
  RedCAP is used to track the enrollment rates to determine the feasibility of a larger randomized controlled trial.
Number of Participants that complete the Intervention as prescribed (Adherence) | During hospitalization, approximately 5 days
  RedCAP is used to track the adherence rates to determine the feasibility of a larger randomized controlled trial.

SECONDARY OUTCOMES:
Duration of Labor (minutes) | Approximately 5 days, length of hospitalization
Mode of Delivery | Approximately 5 days, length of hospitalization
  Vaginal Delivery, Operative Delivery, or Cesarean Section
Number of Postpartum Hemorrhages | Approximately 5 days, length of hospitalization
  Postpartum Hemorrhage as defined as estimated blood loss of over 1000mL.
Number of Treatment Related Adverse Events | Approximately 6 weeks after delivery
Neonatal health (APGAR Score) | Approximately 5 days, length of hospitalization
  APGAR (Activity, Pulse, Grimace, Appearance, Respiration). A normal APGAR score ranges from 8-10. An abnormal score ranges from 0-7. Each scoring indicator can range from 0 to 2 points.
  Activity (Muscle Tone):
  0 Points: Absent
  1. Point: Flexed Limbs
  2. Points: Active
  Pulse:
  0 Points: Absent
  1. Point: <100 beats per minute
  2. Points: >100 beats per minute
  Grimace (Reflex Irritability):
  0 Points: Floppy
  1. Point: Minimal response to stimulation
  2. Points: Prompt response to stumulation
  Appearance (Skin Color):
  0 Points: Blue/Pale
  1. Point: Pink Body, Blue Extremitites
  2. Points: Pink
  Respiration:
  0 Points: Absent
  1. Point: Slow and Irregular
  2. Points: Vigorous Cry
Neonatal health (Cord Blood Gases) | Approximately 5 days, length of hospitalization
  Normal Ranges Arterial pH: 7.20 - 7.30 Venous pH: 7.25 - 7.35 Base Excess: -8 to -2 mmol/L
  Abnormal Ranges pH < 7.0 (Arterial and Venous) Base Excess < -16 mmol/L (Arterial and Venous)
  Abnormal Ranges indicate potential neonatal hypoxia or acidemia.
Maternal Health (Number of Subject who experience PostPartum Fever) | Approximately 5 days, length of hospitalization
Practicality of Administering Calcium Carbonate, as measured by number of subjects who were administered the total prescribed intervention | Approximately 5 days, length of hospitalization
Race | Day 0
  White, Black or African American, Asian, More than One Race/Other, Unknown/Not Reported
Ethnicity | Day 0
  Hispanic, Non-Hispanic, Unknown/Not Reported

CONTACTS AND LOCATIONS:
Overall Officials: Moeun Son, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Intravenous Calcium to Decrease Blood Loss During Intrapartum Cesarean Delivery: A Randomized Controlled Trial. Obstetrics & Gynecology, 143(1), 104-112. — https://doi.org/10.1097/AOG.0000000000005441
- See also: DailyMed-CALCIUM CARBONATE 500MG tablet, chewable. (n.d.) — https://dailymed.nlm.nih.gov/dailymed/drugInfo.cfm?setid=26bba88a-7db2-4cef-b6b9-03183ee85152
- See also: Economy, K. E., & Abuhamad, A. Z. (2001). Calcium channel blockers as tocolytics. Seminars in Perinatology, 25(5), 264-271. — https://doi.org/10.1053/sper.2001.27165
- See also: Association between ionised calcium and severity of postpartum haemorrhage: A retrospective cohort study. British Journal of Anaesthesia — https://doi.org/10.1016/j.bja.2020.11.020
- See also: Fritz, K., Taylor, K., & Parmar, M. (2024). Calcium Carbonate. In StatPearls. StatPearls Publishing. — http://www.ncbi.nlm.nih.gov/books/NBK562303/
- See also: Grier, R. M. (1947). Elective Induction of Labor**Read before the Chicago Gynecological Society, Nov. 15, 1946. American Journal of Obstetrics and Gynecology, 54(3), 511-516. — https://doi.org/10.1016/S0002-9378(16)39418-2
- See also: Luckas, M. J. M., Taggart, M. J., & Wray, S. (1999). Intracellular calcium stores and agonist-induced contractions in isolated human myometrium. American Journal of Obstetrics and Gynecology, 181(2), 468-476. — https://doi.org/10.1016/S0002-9378(99)70580-6
- See also: Monga, M., Campbell, D. F., & Sanborn, B. M. (1999). Oxytocin-stimulated capacitative calcium entry in human myometrial cells. American Journal of Obstetrics and Gynecology, 181(2), 424-429. — https://doi.org/10.1016/S0002-9378(99)70573-9
- See also: Papandreou, L., Chasiotis, G., Seferiadis, K., Thanasoulias, N. C., Dousias, V., Tsanadis, G., & Stefos, T. (2004). Calcium levels during the initiation of labor. European Journal of Obstetrics & Gynecology and Reproductive Biology, 115(1), 17-22. — https://doi.org/10.1016/j.ejogrb.2003.11.032
- See also: Parratt, J., Taggart, M., & Wray, S. (1994). Abolition of contractions in the myometrium by acidification in vitro. The Lancet, 344(8924), 717-718. — https://doi.org/10.1016/S0140-6736(94)92209-8
- See also: Pehlivanoglu, B., Bayrak, S., & Dogan, M. (2013). A close look at the contraction and relaxation of the myometrium; the role of calcium. Journal of the Turkish German Gynecological Association, 14(4), 230-234. — https://doi.org/10.5152/jtgga.2013.67763
- See also: Labor Induction Techniques: Which Is the Best? Obstetrics and Gynecology Clinics — https://doi.org/10.1016/j.ogc.2017.08.011
- See also: The effects of pH change on Ca++ signaling and force in pregnant human myometrium. American Journal of Obstetrics and Gynecology — https://doi.org/10.1067/mob.2003.229
- See also: Medical management of canine and feline dystocia. Theriogenology — https://doi.org/10.1016/j.theriogenology.2008.04.031
- See also: Dysfunctional Labor and Myometrial Lactic Acidosis: Obstetrics & Gynecology — https://doi.org/10.1097/01.AOG.0000118306.82556.43
- See also: The effect of experimentally induced hypocalcaemia on uterine activity at parturition in the ewe. Theriogenology — https://doi.org/10.1016/0093-691X(84)90446-1
- See also: Whelping and Dystocia: Maximizing Success of Medical Management. Topics in Companion Animal Medicine — https://doi.org/10.1053/j.tcam.2018.03.003
- See also: The Myometrium: From Excitation to Contractions and Labour. In H. Hashitani & R. J. Lang (Eds.), Smooth Muscle Spontaneous Activity — https://doi.org/10.1007/978-981-13-5895-1_10